CLINICAL TRIAL: NCT03459833
Title: Glans Penis Augmentation by Hyaluronic Acid for Treatment of Premature Ejaculation: Randomized Controlled Cross-over Trial
Brief Title: Glans Penis Augmentation by Hyaluronic Acid for Treatment of Premature Ejaculation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Wael Ragab, Clinical demonstrator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PE:HA glans augmentation
Record Dates: First submitted 2018-02-12; First posted 2018-03-09 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Premature Ejaculation
Keywords: premature ejaculation; IELT; hyaluronic acid; glans penis augmentation
MeSH Terms: conditions — Premature Ejaculation | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Patients with premature ejaculation according to the definition of Fourth International Consultation on Sexual Medicine 2015
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): 15 patients They will receive a topical anesthetic agent for 30 minutes (Emla cream; lidocaine 25 mg, prilocaine 25 mg, Astra Xeneca, Mississauga, Canada) followed by injection of two prefilled 1 ml syringes with 30 G needle of hyaluronic acid (HA; Teosyal® PureSense Global Action, Teoxane Laboratories, Geneva, Switzerland). After 18 months from the HA injection, cross-over to placebo arm will be done.
  Interventions: Drug: Hyaluronic Acid
- group 2 (Placebo Comparator): They receive by the same method 2 ml saline as a placebo. After one month of the injection, cross-over to HA arm will be done.
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Hyaluronic Acid — Glans penis augmentation using multiple puncture technique as described by Abdallah et al. (2012) with minor modifications. HA is injected at two circular levels: one at the level of corona of glans penis and a second circular level is mid-way between the corona and urethral meatus. Six injections are injected at coronal level and four are injected in the second level, each injection is of 0.2 ml and is injected into deep dermis.

SUMMARY:
This randomized controlled cross-over study aims to evaluate the effect and safety of glans penis augmentation using Hyaluronic acid in the treatment of premature ejaculation in compare with placebo .

ELIGIBILITY:
Inclusion Criteria:

* occurrence of ejaculation in patients with lifelong premature ejaculation (LL PE) within 1 minute form vaginal penetration in all or almost all occasions starting from the first sexual experience, and within 3 minutes in patients with acquired premature ejaculation (A PE), along with inability to delay ejaculation on all or nearly all vaginal penetrations, with negative personal consequences, such as distress, bother, frustration, and/or the avoidance of sexual intimacy

Exclusion Criteria:

* Erectile dysfunction
* Hypo or hyperthyroidism
* Hypogonadism
* Hyperprolactinemia
* Drug abuse
* Psychiatric disorders or related medications

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
IELT | Change from baseline after one month
  Intra-vaginal Ejaculation Latency Time
AIPE | Change from baseline after one month
  Arabic index of premature ejaculation

SECONDARY OUTCOMES:
IELT | Change from baseline after three, six and nine months
  Intra-vaginal Ejaculation Latency Time

CONTACTS AND LOCATIONS:
Overall Officials: Hamed A Hamed, MD, Study Director — Professor of Andrology, Cairo University